CLINICAL TRIAL: NCT05740904
Title: Efficacy and Safety of New Defocus Spectacle Lens in Preventing Progression of Myopia Compared With the Conventional Single-vision Spectacle Lens: a Randomized Controlled Trial Among Chinese Children
Brief Title: Efficacy and Safety of the New Defocus Spectacle Lens in Preventing Progression of Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023KYPJ006
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-03

CONDITIONS: Myopia
Keywords: Defocused lens; Myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New defocus spectacle lens (Experimental): The children in the experimental group will wear new defocus spectacle lens and receive follow-up examinations every half year.
  Interventions: Other: New defocus spectacle lenses
- Conventional aspheric single-vision spectacle lenses (Active Comparator): The children in the control group will wear conventional aspheric single-vision spectacles and receive follow-up examinations every half year.
  Interventions: Other: Convenional aspheric single-vision spectacle lenses

INTERVENTIONS:
Other: New defocus spectacle lenses — The children in the new defocus spectacle lens group will wear new defocus spectacle and receive follow-up examinations every half year.
  Arms: New defocus spectacle lens
Other: Convenional aspheric single-vision spectacle lenses — The children in the convenional aspheric spectacle lenses group will wear conventional aspheric single-vision spectacle and receive follow-up examinations every half year.
  Arms: Conventional aspheric single-vision spectacle lenses

SUMMARY:
The clinical effects of new technical spectacles with refractive correction function are mixed. A randomised trial is designed to compare the effects of new defocusing spectacle lenses and traditional aspheric spectacle lenses on myopia progression in Chinese children aged 6-14 years.

DETAILED DESCRIPTION:
Myopia has become the focus of global attention.

There has been a lot of evidence that soft bifocal contact lenses, corneal plastic lenses, low-concentration atropine and outdoor time can reduce the incidence and progress of myopia, while the clinical effects of new technical spectacles with refractive correction function are mixed. Among the strategies of myopia control through optical intervention, the clinical researches of the bifocal spectacle lens showed that the myopia progression can be slowed by about 50% in two years. However, for active children, wearing 1.50D binoculars may increase the risk of injury caused by falls. Moreover, DIMS (Defocus Incorporated Multiple Segments) spectacle lens which also reported that myopia can be effectively controlled is the effect of reducing the far-sighted defocus of omnidirectional off-axis aberration. Although the DIMS lens do not have the discomfort of wearing like the bifocal lens, because several small defocusing areas divide the imaging, the field of vision will feel uncomfortable vibration, or feel scattered light, which will hinder the field of vision.

Like DIMS lens, defocus spectacle lens aims to suppress hyperopia defocus caused by omni-directional off-axis aberration. The method is to set the focal depth extension area and optical center (refractive correction area) of astigmatism with relatively positive refractive power in the surrounding concentric circle area. The precise focusing position of astigmatism, that is, the defocusing amount of the forward refractive force as the equivalent spherical lens, is about 2.75D as the same as the DIMS lens. The change from the two straight focus lines in the front and back directions of astigmatism to the point image distribution of precise focus is very gentle, so there will be no sharp point image change like the DIMS lens, which can inhibit the discomfort of the field of vision being divided.

This study plans to design a randomised trial to compare the effects of new defocusing spectacle lenses and traditional aspheric spectacle lenses on myopia progression in Chinese children aged 6-14 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 14 years;
* Under the condition of bilateral cycloplegic autorefraction, the spherical refractive error of -1.00 to -3.50 D in each eye and astigmatism of not more than 1.50 D and anisometropia of not more than 1.00 D;
* Best-corrected visual acuity of equal or better than 0.00 LogMAR (>= 1.0 as Snellen).
* The intraocular pressure of 10 to 21mmHg.
* Volunteer to participate in this clinical trial with signature of the informed consent form.

Exclusion Criteria:

* History of eye injury or intraocular surgery;
* Clinically abnormal slit-lamp findings
* Abnormal fundus examination
* Ocular disease, such as uveitis and other inflammatory diseases, glaucoma, cataract, fundus diseases, eye tumors, dominant strabismus, and any eye diseases that affect visual function;
* Systemic diseases causing low immunity (such as diabetes, Down's syndrome, rheumatoid arthritis, psychotic patients or other diseases that researchers think are not suitable for wearing glasses);
* Participation of the drug clinical trial within three month and the device clinical trial within one month;
* Only one eye meets the inclusion criteria;
* Unable to have regular follow-up
* Participation of any myopia control clinical research trial within three months, and currently using rigid contact lenses (including nursing products), multifocal contact lenses, progressive multifocal lenses and other specially designed myopia control lenses, atropine drugs, etc.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Changes of spherical equivalent refraction (SER) at one year | 1 year
  The difference of SER (Diopter) at one year compared with baseline SER. SER will be measured after cycloplegia.

SECONDARY OUTCOMES:
Changes of axial length (AL) at one year | 1 year
  The difference of AL (mm) at one year compared with baseline AL. AL will be measured by IOLMaster-700.
Change of anterior chamber depth (ACD) at one year | 1 year
  The difference of ACD (mm) at one year compared with baseline ACD. ACD will be measured by IOLMaster-700.
Change of lens thickness (LT) at one year | 1 year
  The difference of LT (mm) at one year compared with baseline LT. LT will be measured by IOLMaster-700.
Change of corneal power (CP) at one year | 1 year
  The difference of CP (diopter) at one year compared with baseline CP. CP will be measured by IOLMaster-700.
Best corrected visual acuity（BCVA） at one year | 1 year
  BCVA will be measured at baseline and one year by EDTRS visual acuity chart.
Binocular visual function at one year | 1 year
  Binocular visual function which is a qualitative outcome assessed by a series of tests will be measured every half year.
Choroidal thickness at one year | 1 year
  The difference of Choroidal thickness (μm) at one year compared with baseline measure. Choroidal thickness will be measured by OCTA.
Visual scale score at six months | 6 months
  Visual scale score measured by the Chinese version of the pediatric refractive error profile2 (PREP2) and is scaled from 0 (poor quality of life) to 100 (good quality of life).
Visual scale score at one year | 1 year
  Visual scale score measured by the Chinese version of the pediatric refractive error profile2 (PREP2) is scaled from 0 (poor quality of life) to 100 (good quality of life).
Time length of wearing spectcales at one year | 1 year
  Time length of wearing spectcales will be collected every half year. Participants will report the approximate time of wearing glasses per day and days per week.
Safty of wearing the spectacle lens | 1 year
  Safty of wearing the spectacle lens which is a qualitative outcome will be evaluated every half year by prespecified measures and definations through symptoms and signs, intraocular pressure#slit lamp and ocular fundus checks.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfa Zeng, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Trends in prevalence of blindness and distance and near vision impairment over 30 years: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e130-e143. doi: 10.1016/S2214-109X(20)30425-3. Epub 2020 Dec 1. PMID 33275950
- [Background] Burton MJ, Ramke J, Marques AP, Bourne RRA, Congdon N, Jones I, Ah Tong BAM, Arunga S, Bachani D, Bascaran C, Bastawrous A, Blanchet K, Braithwaite T, Buchan JC, Cairns J, Cama A, Chagunda M, Chuluunkhuu C, Cooper A, Crofts-Lawrence J, Dean WH, Denniston AK, Ehrlich JR, Emerson PM, Evans JR, Frick KD, Friedman DS, Furtado JM, Gichangi MM, Gichuhi S, Gilbert SS, Gurung R, Habtamu E, Holland P, Jonas JB, Keane PA, Keay L, Khanna RC, Khaw PT, Kuper H, Kyari F, Lansingh VC, Mactaggart I, Mafwiri MM, Mathenge W, McCormick I, Morjaria P, Mowatt L, Muirhead D, Murthy GVS, Mwangi N, Patel DB, Peto T, Qureshi BM, Salomao SR, Sarah V, Shilio BR, Solomon AW, Swenor BK, Taylor HR, Wang N, Webson A, West SK, Wong TY, Wormald R, Yasmin S, Yusufu M, Silva JC, Resnikoff S, Ravilla T, Gilbert CE, Foster A, Faal HB. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health. 2021 Apr;9(4):e489-e551. doi: 10.1016/S2214-109X(20)30488-5. Epub 2021 Feb 16. No abstract available. PMID 33607016
- [Background] He M, Xiang F, Zeng Y, Mai J, Chen Q, Zhang J, Smith W, Rose K, Morgan IG. Effect of Time Spent Outdoors at School on the Development of Myopia Among Children in China: A Randomized Clinical Trial. JAMA. 2015 Sep 15;314(11):1142-8. doi: 10.1001/jama.2015.10803. PMID 26372583
- [Background] Hoseini-Yazdi H, Vincent SJ, Read SA, Collins MJ. Astigmatic Defocus Leads to Short-Term Changes in Human Choroidal Thickness. Invest Ophthalmol Vis Sci. 2020 Jul 1;61(8):48. doi: 10.1167/iovs.61.8.48. PMID 32729913
- [Background] Kanda H, Oshika T, Hiraoka T, Hasebe S, Ohno-Matsui K, Ishiko S, Hieda O, Torii H, Varnas SR, Fujikado T. Effect of spectacle lenses designed to reduce relative peripheral hyperopia on myopia progression in Japanese children: a 2-year multicenter randomized controlled trial. Jpn J Ophthalmol. 2018 Sep;62(5):537-543. doi: 10.1007/s10384-018-0616-3. Epub 2018 Aug 6. PMID 30083910
- [Background] Lam CSY, Tang WC, Tse DY, Lee RPK, Chun RKM, Hasegawa K, Qi H, Hatanaka T, To CH. Defocus Incorporated Multiple Segments (DIMS) spectacle lenses slow myopia progression: a 2-year randomised clinical trial. Br J Ophthalmol. 2020 Mar;104(3):363-368. doi: 10.1136/bjophthalmol-2018-313739. Epub 2019 May 29. PMID 31142465
- [Background] Yam JC, Zhang XJ, Zhang Y, Wang YM, Tang SM, Li FF, Kam KW, Ko ST, Yip BHK, Young AL, Tham CC, Chen LJ, Pang CP. Three-Year Clinical Trial of Low-Concentration Atropine for Myopia Progression (LAMP) Study: Continued Versus Washout: Phase 3 Report. Ophthalmology. 2022 Mar;129(3):308-321. doi: 10.1016/j.ophtha.2021.10.002. Epub 2021 Oct 7. PMID 34627809
- [Background] Zhang HY, Lam CSY, Tang WC, Leung M, To CH. Defocus Incorporated Multiple Segments Spectacle Lenses Changed the Relative Peripheral Refraction: A 2-Year Randomized Clinical Trial. Invest Ophthalmol Vis Sci. 2020 May 11;61(5):53. doi: 10.1167/iovs.61.5.53. PMID 32460315